CLINICAL TRIAL: NCT06080230
Title: The Effect of Resilience Psychoeducation Program Based on Positive Psychotherapy on Nurses Resilience and Balanced Life Skills
Brief Title: The Effect of Resilience Psychoeducation Program Based on Positive Psychotherapy on Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duzce University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DuzceUsedaoner081081
Record Dates: First submitted 2023-04-27; First posted 2023-10-12 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2023-10

CONDITIONS: Psychological Stress
Keywords: Psychoeducation Program; Nurses; Adult resillience scale
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychoeducation Program Group (Active Comparator): Participants in the 8-week Program
  Interventions: Behavioral: Participants in the 8-week program
- Control Group (No Intervention): Those who do not participate in the 8-week Program

INTERVENTIONS:
Behavioral: Participants in the 8-week program — Psychological resilience program based on positive psychotherapy was applied to nurses
  Arms: Psychoeducation Program Group

SUMMARY:
The Effect of Resilience Psychoeducation Program Based on Positive Psychotherapy on Nurses

DETAILED DESCRIPTION:
Based on the principles of positive psychology, Positive Psychotherapy integrates symptoms with strengths, resources with risks, weaknesses with values, and hopes with regret to understand the natural complexities of human experiences in a balanced way. This includes cognitive restructuring of the individual, reviewing expectations, and acquiring new goals.

Resilience is a person's process of adapting, resilience, or the ability to successfully cope with change/disaster against major stressors such as a trauma, a threat, a tragedy, or familial and relational distress, serious health problems, workplace and financial problems. It is stated that people with high psychological resilience are more successful in adapting to change and struggling against obstacles, and people with high psychological resilience experience less emotional exhaustion.10 Possible risky situations that individuals encounter in their work life and the protective factors they have also affect their psychological resilience. It is also stated that psychological resilience is an important concept for nurses who are faced with many risk factors, especially in business life, and who have to provide professional care to patients who are in difficult situations and in need, and who have to comfort the patient.1 The effectiveness of developing and strengthening psychological resilience in coping with the stressful environment of nursing has been proven. It is stated that among the coping resources of nurses, adequate rest, self-care and social support are of great importance and that these resources are positively related to the quality of life.

The aim of this research is to determine the effect of the Psychological Resilience Psychoeducation Program Based on Positive Psychotherapy on the resilience of nurses and to determine their balanced life skills.

ELIGIBILITY:
Inclusion Criteria:

* Working as a nurse at Düzce University Health Application and Research Center
* Individuals who voluntarily agree to participate in the research will be included.

Exclusion Criteria:

* The acute phase of a psychiatric illness

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Resilience Scale for Adults scores | 8 weeks
  Effect of Psychoeducation Program on nurse adult resilience scale scores.In order to avoid biased evaluations in choosing the items, the scale uses a format in which the positive and negative features are on different sides and there are five separate boxes for the answers. In the schematic evaluation, the scoring method is free for measuring psychological resilience as high or low.

CONTACTS AND LOCATIONS:
Locations (1):
- Duzce University, Merkez, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No